CLINICAL TRIAL: NCT02006706
Title: An Open-label Study to Evaluate the Effect of MabThera in Combination With Methotrexate on Disease Activity in Patients With Active Rheumatoid Arthritis After DMARD Treatment Failure
Brief Title: A Study of MabThera/Rituxan (Rituximab) in Combination With Methotrexate in Patients With Rheumatoid Arthritis and Inadequate Response to DMARD Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML20388
Record Dates: First submitted 2013-12-05; First posted 2013-12-10 (Estimated); Results first posted 2014-11-06 (Estimated); Last update posted 2017-08-21 (Actual); Status verified 2017-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab; Methotrexate; Methylprednisolone

ARMS (1):
- MabThera/Rituxan (Experimental)
  Interventions: Drug: rituximab [MabThera/Rituxan]; Drug: methotrexate; Drug: methylprednisolone

INTERVENTIONS:
Drug: rituximab [MabThera/Rituxan] — 1000 mg iv Days 1 and 15
Drug: methotrexate — 10 - 25 mg/week
Drug: methylprednisolone — iv administration on Day 1 and 15 prior to MabThera/Rituxan infusion

SUMMARY:
This study will evaluate the efficacy and safety of MabThera/Rituxan plus methotrexate in patients with active rheumatoid arthritis who have had an inadequate response to at least 1 DMARD treatment. All patients will receive MabThera (1000mg iv infusion) on days 1 and 15, and methotrexate (10-25mg po) weekly. The anticipated time on study treatment is 3-12 months.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-80 years of age;
* rheumatoid arthritis after inadequate response to >=1 DMARD treatment;
* active disease;
* DMARDs other than methotrexate withdrawn for at least 4 weeks prior to start of study treatment.

Exclusion Criteria:

* autoimmune disease other than rheumatoid arthritis;
* bone/joint surgery within 8 weeks prior to screening, or joint surgery planned within 24 weeks of MabThera infusion;
* concurrent treatment with any DMARD or antiTNF-alfa;
* intra-articular or parenteral corticosteroids within 4 weeks prior to screening.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2006-08-10 (Actual); Primary Completion 2007-11-23 (Actual); Study Completion 2007-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- Serbia (3):
  - Belgrade
  - Niška Banja
  - Nova Sad

RESULTS

PARTICIPANT FLOW:
Groups:
- Rituximab/Methylprednisolone/Methotrexate (MTX): Participants received rituximab 1000 milligrams (mg), intravaneously (IV), and methylprednisolone 100 mg, IV, on Days 1 and 15. Participants also received MTX, 10 to 25 mg per week (at a stable dose at the discretion of investigator and in accordance with the local label), orally (or parenterally, as prescribed) and folate 5 mg per week, orally, for up to 24 weeks.
Period: Overall Study
Arm/Group | Rituximab/Methylprednisolone/Methotrexate (MTX)
Started | 15
Completed | 14
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Per-protocol (PP) population: The 14 enrolled participants who were compliant with the protocol and not lost to follow-up.
Groups:
- Rituximab/Methylprednisolone/MTX: Participants received rituximab 1000 mg, IV, and methylprednisolone 100 mg, IV, on Days 1 and 15. Participants also received MTX, 10 to 25 mg per week (at a stable dose at the discretion of investigator and in accordance with the local label), orally (or parenterally, as prescribed) and folate 5 mg per week, orally, for up to 24 weeks.
Arm/Group | Rituximab/Methylprednisolone/MTX
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.29 (11.89)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Serbia | 14

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Disease Activity Score Based on 28-Joint Count (DAS28) at Week 24
Description: DAS28 was calculated from the number of swollen joints and painful joints using the 28 joints count, the erythrocyte sedimentation rate (ESR) (millimeters per hour [mm/hour]) and patient's global assessment (PGA) of disease activity (participant-rated arthritis activity assessment using visual analog scale [VAS]) with transformed scores ranging 0 to 10; higher scores indicated greater affectation due to disease activity). DAS28 less than or equal to (≤)3.2 equals (=) low disease activity, DAS28 greater than (>)3.2 to 5.1 = moderate to high disease activity.
Time Frame: Baseline, Week 24
Population: Per Protocol (PP) Population: included all participants who received at least one dose of study drug and who did not have any protocol violations.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rituximab/Methylprednisolone/MTX
Number analyzed (Participants) | 14
score on a scale | 2.98 (1.80)
Statistical Analysis 1: Comparison: Rituximab/Methylprednisolone/MTX; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = 2.98, 95% CI 2-sided [1.73 to 4.22], Standard Error of Mean 0.606 — The null hypothesis was that there was no difference between the DAS28 at baseline and DAS28 after 24 weeks of follow-up

2. Secondary Outcome: Health Assessment Questionnaire-Disability Index (HAQ-DI)
Description: HAQ-DI: participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week. Each item scored on 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0 = least difficulty and 3 = extreme difficulty.
Time Frame: Baseline, Week 24
Population: PP Population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rituximab/Methylprednisolone/MTX
Number analyzed (Participants) | 14
score on a scale
  Baseline | 1.91 (0.687)
  Week 24 | 1.05 (0.960)
Statistical Analysis 1: Comparison: Rituximab/Methylprednisolone/MTX; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were reported starting with the first dose of study drug through the end of the study (24 weeks total).
Arm/Group | Rituximab/Methylprednisolone/MTX
Serious Adverse Events (participants affected / at risk) | 2/14
Other Adverse Events (participants affected / at risk) | 0/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab/Methylprednisolone/MTX (N=14)
Infarctus myocardii (Cardiac disorders) | 1
Enterocolitis acuta (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request the Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.